CLINICAL TRIAL: NCT04949594
Title: Relief of Pain in Patients With Cervical Dystonia Through the Use of Sensory Threshold TENS
Brief Title: Relief of Pain in Patients With Cervical Dystonia Through the Use of Transcutaneous Electric Nerve Stimulation (TENS)
Acronym: TENDYS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI213
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Cervical Dystonia; Pain
Keywords: cervical dystonia; pain; TENS
MeSH Terms: conditions — Torticollis; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TENS — application on muscles where pain is situated (cervical)
  Other Names: transcutaneous electrical nerve stimulation

SUMMARY:
Dystonia is a chronic neurological condition that impacts the quality of life due to decreased mobility, social repercussions caused by others's perception of abnormal involuntary movement and frequent pain. Botulinum toxin has been shown to be effective in reducing pain in dystonia. However, many patients remain painful despite the injections, especially when the decrease in the effect of the latter, performed every 3 months on average. Despite frequent use of TENS in pain relief, only a few small studies studying TENS in dystonia were published and none of them reported TENS effects on dystonic pain using sensory threshold.

This study aimed to quantify the efficacy and tolerance of TENS in the indication of pain related to dystonia, focusing on cervical dystonia which is the most common form of dystonia.

DETAILED DESCRIPTION:
TENDYS (TENs use in cervical DYStonia) is an observational, prospective, single arm, monocentric study including subjects between September 2019 and July 2020 with cervical dystonia treated or not with botulinum neurotoxin (BoNT) type A at the Nancy Regional University Hospital.

All patients who benefited from a simple follow-up or injections of BoNT every 3 or 4 months for a painful cervical dystonia were proposed the use of TENS during a neurologic consultation with one of two specialist physicians trained to cervical dystonia. Patients who accepted had to give informed consent and were re-evaluated about 1 month later to ensure that pain persisted and to have a demo of TENS. The electro-stimulator was delivered to posterior cervical muscles over or close to the painful site, according to a Conventional or High frequency/Low intensity mode (Gate control). Patients were encouraged to use the machine daily, as often and long and possible, except for sleeping and driving.

Follow-up assessments of pain occurred at the consultation toxin injection 3 months later and at 4 months for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient having received complete information on the organization of the research and not having objected to the exploitation of the data
* patient admitted to neurology consultation for cervical dystonia treated with botulinum toxin

Exclusion Criteria:

* Patient under legal protection
* Minor patient
* Patient refusing to give consent
* Patient with exclusive radicular or truncal involvement
* Missing data or absence of established reactogenic threshold

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient admitted to a neurology consultation for cervical dystonia treated with botulinum toxin.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Mean change of Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Total score | 3 months
  Toronto Western Spasmodic Torticollis Rating Scale (abbreviated TWSTRS) is a mixed clinician and patient rated cervical dystonia-specific scale. TWSTRS total score is scored from 0-85 (best to worst).

SECONDARY OUTCOMES:
Mean change of Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Severity, -Disability and -Pain subscores | 3 months
  The TWSTRS is comprised of 3 subscales : severity (range 0-35), disability (range 0-30), and pain (range 0-20), each of which is scored independently (best to worst).
Mean change of Pain Numeric Rating Scale score | 3 months
  Pain Numeric Rating Scale (abbreviated PNRS) is ranking 0-10, with 0 meaning "No pain" and 10 meaning "Pain as bad as you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: SOLENE FRISMAND-KRYLOFF, Principal Investigator — CHRU Nancy
Locations (1):
- Frismand-Kryloff, Nancy, France

IPD SHARING:
Plan to Share IPD: No